CLINICAL TRIAL: NCT02151513
Title: Pilot Study on the Effect of Intrathecal Opioids on Immune Function in Humans With Cancer Pain
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Shane Brogan, Associate Professor, Anesthesiology, University of Utah
Other Study IDs: IRB_00057738
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Cancer-associated Pain
Keywords: Cancer-associated pain; Immune function
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Pain: Placement of an intrathecal pump
  Interventions: Device: Intrathecal Pump Placement

INTERVENTIONS:
Device: Intrathecal Pump Placement
  Other Names: Medtronic SyncroMed II

SUMMARY:
The purpose of this study is to examine the changes in immune function, as measured by biomarkers in the blood, that happen with intrathecal (spinal) delivery of opioid medications for the treatment of moderate to severe cancer pain.

Hypothesis: Treatment of pain with intrathecal (spinal) therapy is associated with little alteration of immune function as measured by biomarkers in the blood of cancer patients with moderate to severe pain.

DETAILED DESCRIPTION:
Biomarkers of immune function will be measured before and after patients receive an intrathecal pain pump for management of cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Evaluation by a pain management physician and confirmation that cancer is the primary etiology of patient's pain
* Moderate to severe pain, as specified by a baseline Pain Rating Score of 5 or above on a scale from 0 (no pain) to 10 (worst pain imaginable) despite current opioid therapy
* Pain management plan (as developed by Interventional Pain Service, patient and primary service) that includes placement of an intrathecal drug delivery system for pain management
* Able and willing to give informed consent

Exclusion Criteria:

* Patients with an expected life expectancy of less than 12 weeks
* Patients not felt be a safe surgical candidate by pain management physician for placement of and intrathecal drug delivery system (IDDS) due to the presence of severe medical comorbidities
* Patients who are not a candidate for intrathecal drug therapy due to coagulopathy, concurrent necessary use of blood thinners, presence of systemic infection, drug allergy to analgesic agent, evidence of CSF obstruction or other technical factor
* Severe or untreated psychiatric disease
* Refusal of informed consent
* Pregnant patients or patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer-associated pain who are receiving an intrathecal pump for management of cancer pain
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in biomarker values | Before, 4 weeks after and 8 weeks after intrathecal pump placement
  Change in biomarker values as measured by blood

SECONDARY OUTCOMES:
Change in Quality of Life as measured by a Brief Pain Inventory | Before, 4 weeks after and 8 weeks after intrathecal pump placement
  Quality of life surveys as measured by a Brief Pain Inventory questionnaire
Change in Quality of Life as measured by MD Anderson Symptom Inventory | Before, 4 weeks after and 8 weeks after intrathecal pump placement
  Quality of life surveys as measured by MD Anderson Symptom Inventory questionnaire
Serum Opioid Levels | Before, 4 weeks after and 8 weeks after intrathecal pump placement
  Serum Opioid Levels

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Hosptial, Salt Lake City, Utah, United States